CLINICAL TRIAL: NCT02287896
Title: Pharmacokinetics and Safety of Roledumab, a Fully Human Recombinant Monoclonal Anti-RhD Antibody, in RhD-negative Pregnant Woman Carrying an RhD-positive Foetus: a Phase IIb, Multicenter, Open-label Study
Brief Title: Pharmacokinetics and Safety of Roledumab in RhD-negative Pregnant Women Carrying an RhD-positive Foetus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ADNC-1301; 2013-000269-35 (EudraCT Number)
Record Dates: First submitted 2014-10-28; First posted 2014-11-11 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2019-08

CONDITIONS: Rh Disease
Keywords: RhD-negative pregnant woman; anti-RhD antibody
MeSH Terms: interventions — LFB-R593

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roledumab Open-label IM (Experimental): - Planned antenatal prophylaxis: A single dose of 300 µg IM of Roledumab at 28 or 29 weeks of gestation.
  - Antenatal prophylaxis following sensitizing events: One or more dose(s) of 300μg IM anti-RhD antibodies (Rhophylac or Roledumab) based on the Kleihauer-test as soon as possible and no later than 72 hours after event occurrence.
  - Postnatal prophylaxis: Roledumab should be administered to the mother as soon as possible within 72 hours of delivery of an RhD positive infant.
  The postnatal dose must still be given even when antenatal prophylaxis has been administered.
  Before Roledumab 300μg IM postnatal administration, a Kleihauer-Betke test will be performed on maternal blood sample taken no earlier than 30 min after delivery in order to determine the volume of foetomaternal hemorrhage (FMH).
  Interventions: Drug: ROLEDUMAB
- Roledumab Open-label IV (Experimental): - Planned antenatal prophylaxis: A single dose of 300 µg IV of Roledumab at 28 or 29 weeks of gestation.
  - Antenatal prophylaxis following sensitizing events: One or more dose(s) of 300μg IV anti-RhD antibodies (Rhophylac or Roledumab) based on the Kleihauer-test as soon as possible and no later than 72 hours after event occurrence.
  - Postnatal prophylaxis: Roledumab should be administered to the mother as soon as possible within 72 hours of delivery of an RhD positive infant.
  The postnatal dose must still be given even when antenatal prophylaxis has been administered.
  Before Roledumab 300μg IV postnatal administration, a Kleihauer-Betke test will be performed on maternal blood sample taken no earlier than 30 min after delivery in order to determine the volume of foetomaternal hemorrhage (FMH).
  Interventions: Drug: ROLEDUMAB

INTERVENTIONS:
Drug: ROLEDUMAB — See Arm description
  Other Names: LFB-R593

SUMMARY:
The aim of this study is to assess the pharmacokinetic profile of Roledumab 300μg IM / IV in RhD-negative pregnant women carrying an RhD-positive foetus.

To assess the safety of Roledumab in RhD-negative pregnant women and in RhD-positive fetus and newborns.

In addition the efficacy of Roledumab 300μg IM and IV to prevent RhD alloimmunisation in RhD-negative pregnant women carrying an RhD-positive fetus and the immunogenicity of Roledumab will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form provided by the subject prior to proceeding with any study-related procedure,
* At least 18 years old,
* Pregnancy between 12 and 27 weeks gestational age as confirmed by early ultrasound,
* Pregnant RhD-negative woman carrying an RhD-positive fetus confirmed by a non-invasive fetal RhD genotyping test,
* Negative serology: HIV (1 and 2), hepatitis C and hepatitis B, except for positive results due to vaccinations,
* Covered by healthcare insurance in accordance with local requirements.

Exclusion Criteria:

* RhD allo-immunized subject,
* Positive for ADA test,
* Multiple fetuses,
* Occurrence of a documented potential sensitizing event in this pregnancy before the antenatal IMP administration,
* Prior administration of anti-RhD immunoglobulin during the current pregnancy,
* Known clinically relevant maternal or fetal abnormality (e.g., as determined by ultrasound or genetic testing), such as placenta previa,
* History of anaphylactic or severe systemic reaction to immunoglobulin of any origin,
* Current diagnosis of an immune disease which by itself or its treatment could impair the safety and/or efficacy evaluation of Roledumab in this study. These diseases are: All immune deficiencies, particularly those requiring IV-Ig supplementation or other systemic treatment / connective tissue and autoimmune diseases (e.g., systemic lupus erythematosus, antiphospholipid syndrome, Sjögren's syndrome, rheumatoid arthritis, ankylosing spondylarthritis) requiring systemic immunosuppressive treatment / allergic and inflammatory diseases requiring systemic immunosuppressive treatment,
* Clinically significant medical history contraindicating the participation in the study according to the judgment of the Investigator or Sponsor,
* Clinically significant laboratory (hematology, blood chemistry, or urinalysis) parameters,
* For the IM arm only, subject with coagulation disorders contraindicating intramuscular injection (patient will still be considered for the IV arm),
* Transfusion of RhD-positive blood or blood derived products within the 6 months prior to enrolment,
* Anticipated poor compliance with the study procedures,
* Subject within exclusion period further to her participation in a clinical study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-04; Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert WINER, MD, Principal Investigator — Nantes University Hospital
Locations (8):
- France (8):
  - Jeanne de Flandre Hospital, Lille
  - Croix-Rousse Maternity, Lyon
  - University Hospital Center, Nantes
  - Armand-Trousseau Hospital, Paris
  - Port-Royal Maternity, Paris
  - Poissy-Saint-Germain-en-Laye Hospital, Poissy
  - Maison Blanche Hospital, Reims
  - Paule de Viguier Hospital, Toulouse

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 100 subjects were pre-screened in the pre-assigment period, only 62 subjects were included in the study.
Groups:
- IM Arm Roledumab: Roledumab Open-label IM
  * Planned antenatal prophylaxis: A single dose of 300 µg IM of Roledumab at 28 or 29 weeks of gestation.
  * Antenatal prophylaxis following sensitizing events: One or more dose(s) of 300μg IM anti-RhD antibodies (Rhophylac or Roledumab) based on the Kleihauer-test as soon as possible and no later than 72 hours after event occurrence.
  * Postnatal prophylaxis: Roledumab should be administered to the mother as soon as possible within 72 hours of delivery of an RhD positive infant.
  The postnatal dose must still be given even when antenatal prophylaxis has been administered.
  Before Roledumab 300μg IM postnatal administration, a Kleihauer-Betke test will be performed on maternal blood sample taken no earlier than 30 min after delivery in order to determine the volume of foetomaternal hemorrhage
- IV Arm Roledumab: Roledumab Open-label IV
  * Planned antenatal prophylaxis: A single dose of 300 µg IV of Roledumab at 28 or 29 weeks of gestation.
  * Antenatal prophylaxis following sensitizing events: One or more dose(s) of 300μg IV anti-RhD antibodies (Rhophylac or Roledumab) based on the Kleihauer-test as soon as possible and no later than 72 hours after event occurrence.
  * Postnatal prophylaxis: Roledumab should be administered to the mother as soon as possible within 72 hours of delivery of an RhD positive infant.
  The postnatal dose must still be given even when antenatal prophylaxis has been administered.
  Before Roledumab 300μg IV postnatal administration, a Kleihauer-Betke test will be performed on maternal blood sample taken no earlier than 30 min after delivery in order to determine the volume of foetomaternal hemorrhage.
Period: Screening Visit V1
Arm/Group | IM Arm Roledumab | IV Arm Roledumab
Started | 36 | 26
Completed | 36 | 26
Not Completed | 0 | 0
Period: First Injection Visit
Arm/Group | IM Arm Roledumab | IV Arm Roledumab
Started | 36 | 26
Completed | 36 | 26
Not Completed | 0 | 0
Period: Second Injection Visit
Arm/Group | IM Arm Roledumab | IV Arm Roledumab
Started | 36 | 26
Completed | 36 | 25
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- IM Arm Roledumab: Roledumab Open-label IM
  Dosage and frequency of administration:
  * Planned antenatal prophylaxis: A single dose of 300 µg IM of Roledumab at 28 or 29 weeks of gestation.
  * Antenatal prophylaxis following sensitizing events: One or more dose(s) of 300μg IM anti-RhD antibodies (Rhophylac or Roledumab) based on the Kleihauer-test as soon as possible and no later than 72 hours after event occurrence.
  * Postnatal prophylaxis: Roledumab should be administered to the mother as soon as possible within 72 hours of delivery of an RhD positive infant.
  The postnatal dose must still be given even when antenatal prophylaxis has been administered.
  Before Roledumab 300μg IM postnatal administration, a Kleihauer-Betke test will be performed on maternal blood sample taken no earlier than 30 min after delivery in order to determine the volume of foetomaternal hemorrhage
- IV Arm Roledumab: Roledumab Open-label IV
  Dosage and frequency of administration:
  * Planned antenatal prophylaxis: A single dose of 300 µg IV of Roledumab at 28 or 29 weeks of gestation.
  * Antenatal prophylaxis following sensitizing events: One or more dose(s) of 300μg IV anti-RhD antibodies (Rhophylac or Roledumab) based on the Kleihauer-test as soon as possible and no later than 72 hours after event occurrence.
  * Postnatal prophylaxis: Roledumab should be administered to the mother as soon as possible within 72 hours of delivery of an RhD positive infant.
  The postnatal dose must still be given even when antenatal prophylaxis has been administered.
  Before Roledumab 300μg IV postnatal administration, a Kleihauer-Betke test will be performed on maternal blood sample taken no earlier than 30 min after delivery in order to determine the volume of foetomaternal hemorrhage.
- Total: Total of all reporting groups
Arm/Group | IM Arm Roledumab | IV Arm Roledumab | Total
Number analyzed (Participants) | 36 | 26 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 26 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 31.0 [20 to 45] | 31.5 [19 to 41] | 31.0 [19 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 26 | 62
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 36 | 26 | 62

OUTCOME MEASURES:

1. Primary Outcome: CL/F : Apparent Clearance
Description: The parameter was estimated through a population pharmacokinetic model, during which concentration data (ante- and postnatal) obtained after single IM or IV route dose of roledumab.
  All samples (ante- and postnatal samples for IM and IV route) will be used for population PK modeling.
Time Frame: IM: Antenatal PK time points at T0, 48h, 120h, 9d, 29d,59d and Posnatal PK time points at TO, 3d,9d, 6 weeks IV: antenal PK time points at T0, 1h, 24h, 48h, 96-120h, 29d, 59d and Postnatal PK time points at T0, 3d, 9d, 6 weeks.
Measure: Mean (Standard Error); unit: L/h
Groups:
- Population PK (PKS1): Single dose of Roledumab 300 μg has been administered for ante- and postnatal periods.
Arm/Group | Population PK (PKS1)
Number analyzed (Participants) | 60
L/h | 0.0106 (5.91)

2. Primary Outcome: V2/F : Central Volume of Distribution
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Population PK (PKS1)
Number analyzed (Participants) | 60
L | 4.02 (4.98)

3. Primary Outcome: t 1/2 : Terminal Half-life
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: hour
Arm/Group | Population PK (PKS1)
Number analyzed (Participants) | 60
hour | 481.7 (0)

4. Primary Outcome: C Max
Description: C max (maximum observed serum concentration) of Roledumab in all ITT subjects enrolled in the IM arm or the IV arm, who had at least one valid PK assessment after the first IMP administration, providing at least one evaluable PK parameter.
  Only samples post-first administration (antenatal samples) will be analyzed by NCA PK analysis for each study arm.
Time Frame: for IM:T0, 48h, 120h, 9 days, 29 days, 59 days and for IV T0, 1h, 24h, 48h, 96-120h, 29 days, 59 days
Population: In the IV arm (PKS3), the overall number of participants analyzed was 25. Due to a sensitizing event at late stage of pregnancy in one woman and a premature delivery in another woman, the number of subjects in the analyzed population was 23.
Measure: Median (Full Range); unit: ng/mL
Groups:
- IM Arm Roledumab: Arm with RhD-negative pregnant women who were allocated to the IM route of administration of Roledumab.
  - Planned antenatal prophylaxis: A single dose of 300 µg IM of Roledumab at 28 or 29 weeks of gestation.
- IV Arm Roledumab: Arm with RhD-negative women who were allocated to the IV route of administration of Roledumab.
  - Planned antenatal prophylaxis: A single dose of 300 µg IV of Roledumab at 28 or 29 weeks of gestation.
Arm/Group | IM Arm Roledumab | IV Arm Roledumab
Number analyzed (Participants) | 34 | 23
ng/mL | 21.6 [7.98 to 31.5] | 71.8 [42.9 to 91.5]

5. Primary Outcome: T Max
Description: T max (time of the maximum observed plasma concentration) of Roledumab in all ITT subjects enrolled in the IM arm or the IV arm, who had at least one valid PK assessment after the first IMP administration, providing at least one evaluable PK parameter.
  Only samples post-first administration (antenatal samples) will be analyzed by NCA PK analysis for each study arm.
Time Frame: for IM:T0, 48h, 120h, 9 days, 29 days, 59 days and for IV T0, 1h, 24h, 48h, 96-120h, 29 days, 59 days
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Groups:
- IV Arm Roledumab: Arm with RhD-negative women who were allocated to the IV route of administration of Roledumab.
  Planned antenatal prophylaxis: A single dose of 300 µg IV of Roledumab at 28 or 29 weeks of gestation.
Arm/Group | IM Arm Roledumab | IV Arm Roledumab
Number analyzed (Participants) | 34 | 23
hour | 167.21 [46.25 to 671.58] | 1.00 [0.95 to 1.50]

6. Primary Outcome: T 1/2
Description: T 1/2 (apparent plasma terminal elimination half-life) of Roledumab in all ITT subjects enrolled in the IM arm or the IV arm, who had at least one valid PK assessment after the first IMP administration, providing at least one evaluable PK parameter.
  Only samples post-first administration (antenatal samples) will be analyzed by NCA PK analysis for each study arm.
Time Frame: for IM:T0, 48h, 120h, 9 days, 29 days, 59 days and for IV: T0, 1h, 24h, 48h, 96-120h, 29 days, 59 days
Population: In the IM arm, the number of participants analyzed was 34, but only 28 subjects with AUCextrap <30% were eligible.
  In the IV arm, the number of participants analyzed was 25. Due to a sensitizing event at late stage of pregnancy in one woman and a premature delivery in another woman, the number of subjects in the analyzed population was 23.
Measure: Median (Full Range); unit: hour
Arm/Group | IM Arm Roledumab | IV Arm Roledumab
Number analyzed (Participants) | 28 | 23
hour | 462 [379 to 835] | 412 [304 to 748]

7. Primary Outcome: AUC 0-t
Description: AUC 0-t (area under the concentration-time curve from time 0 to time Tlast) of Roledumab in all ITT subjects enrolled in the IM arm or the IV arm, who had at least one valid PK assessment after the first IMP administration, providing at least one evaluable PK parameter.
  Only samples post-first administration (antenatal samples) will be analyzed by NCA PK analysis for each study arm.
Time Frame: for IM: T0, 48h, 120h, 9 days, 29 days, 59 days and for IV T0, 1h, 24h, 48h, 96-120h, 29 days, 59 days
Population: In the IV arm, the number of participants analyzed was 25. Due to a sensitizing event at late stage of pregnancy in one woman and a premature delivery in another woman, the number of subjects in the analyzed population was 23.
Measure: Median (Full Range); unit: h*ng/mL
Groups:
- IM Arm Roledumab: Arm with RhD-negative pregnant women who were allocated to the IM route of administration of Roledumab.
  * Planned antenatal prophylaxis: A single dose of 300 µg IM of Roledumab at 28 or 29 weeks of gestation.
- IV Arm Roledumab: Arm with RhD-negative pregnant women who were allocated to the IV route of administration of Roledumab.
  * Planned antenatal prophylaxis: A single dose of 300 µg IV of Roledumab at 28 or 29 weeks of gestation.
Arm/Group | IM Arm Roledumab | IV Arm Roledumab
Number analyzed (Participants) | 34 | 23
h*ng/mL | 16600 [9450 to 25300] | 24900 [14300 to 38500]

ADVERSE EVENTS:
Time Frame: The safety of roledumab was assessed by recording all AEs occurring during the study, i.e. after signature of the informed consent and until the end of the study. AEs in both mother and fetus/newborn were collected and recorded. The safety of roledumab was to be assessed during the third trimester of pregnancy and during the postnatal follow-up visits up to 12 months after delivery.
Groups:
- IM Arm Roledumab: Arm with RhD-negative pregnant women who were allocated to the IM route of administration of LFB-R593
  Dosage and frequency of administration:
  * Planned antenatal prophylaxis: A single dose of 300 µg IM of Roledumab at 28 or 29 weeks of gestation.
  * Antenatal prophylaxis following sensitizing events: One or more dose(s) of 300μg IM anti-RhD antibodies (Rhophylac or Roledumab) based on the Kleihauer-test as soon as possible and no later than 72 hours after event occurrence.
  * Postnatal prophylaxis: Roledumab should be administered to the mother as soon as possible within 72 hours of delivery of an RhD positive infant.
  The postnatal dose must still be given even when antenatal prophylaxis has been administered.
  Before Roledumab 300μg IM postnatal administration, a Kleihauer-Betke test will be performed on maternal blood sample taken no earlier than 30 min after delivery in order to determine the volume of foetomaternal hemorrhage
- IV Arm Roledumab: Arm with RhD-negative pregnant women who were allocated to the IV route of administration of LFB-R593
  Dosage and frequency of administration:
  * Planned antenatal prophylaxis: A single dose of 300 µg IV of Roledumab at 28 or 29 weeks of gestation.
  * Antenatal prophylaxis following sensitizing events: One or more dose(s) of 300μg IV anti-RhD antibodies (Rhophylac or Roledumab) based on the Kleihauer-test as soon as possible and no later than 72 hours after event occurrence.
  * Postnatal prophylaxis: Roledumab should be administered to the mother as soon as possible within 72 hours of delivery of an RhD positive infant.
  The postnatal dose must still be given even when antenatal prophylaxis has been administered.
  Before Roledumab 300μg IV postnatal administration, a Kleihauer-Betke test will be performed on maternal blood sample taken no earlier than 30 min after delivery in order to determine the volume of foetomaternal hemorrhage.
- All Patients: Arm with RhD-negative pregnant women who were allocated to the IV and the IM route of administration of LFB-R593
Arm/Group | IM Arm Roledumab | IV Arm Roledumab | All Patients
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/26 | 0/62
Serious Adverse Events (participants affected / at risk) | 15/36 | 9/26 | 24/62
Other Adverse Events (participants affected / at risk) | 36/36 | 26/26 | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IM Arm Roledumab (N=36) | IV Arm Roledumab (N=26) | All Patients (N=62)
Abdominal injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Foetal heart rate disorder (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Poland's syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1) — Event diagnosed during pregnancy for the fetus and confirmed in the newborn
Polydactyly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 3 (3)
preterm premature rupture of mebranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 2 (2)
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
Retained placenta of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
premature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 2 (2)
HELLP sydrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
fever neonatal (General disorders) | 2 (2) | 0 (0) | 2 (2)
Pyelocaliectasis (General disorders) | 1 (1) | 0 (0) | 1 (1) — Event diagnosed during pregnacy for the fetus and confirmed in the newborn
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Amniotic cavity infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Neonatal infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IM Arm Roledumab (N=36) | IV Arm Roledumab (N=26) | All Patients (N=62)
C reactive protein increased (Investigations) | 4 (4) | 1 (1) | 5 (5)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 11 (11) | 5 (7) | 16 (18)
Headache (Nervous system disorders) | 11 (16) | 6 (8) | 17 (24)
Afterbirth pain (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 10 (10) | 20 (20)
prolonged labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 5 (5)
prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 4 (4)
Uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1) | 5 (5)
uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4) | 7 (7)
caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1) | 5 (5)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) | 5 (5)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 4 (4) | 4 (4)
Asthenia (General disorders) | 4 (4) | 3 (3) | 7 (7)
Vessel puncture site haematoma (General disorders) | 0 (0) | 4 (4) | 4 (4)
Injection site haematoma (General disorders) | 0 (0) | 8 (8) | 8 (8)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (6) | 12 (13)
Haemorrhoids (Gastrointestinal disorders) | 6 (6) | 9 (10) | 15 (16)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 7 (7) | 10 (10) — 6 mothers and 4 newborns
Infantile colic (Gastrointestinal disorders) | 3 (3) | 3 (3) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Nipple disorder (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 5 (5)
ligament pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (3) | 7 (7)
nasopharyngitis (Infections and infestations) | 6 (6) | 5 (6) | 11 (12)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 4 (4) | 7 (7)
Neonatal candida infection (Infections and infestations) | 4 (4) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT02287896/Prot_002.pdf
  • Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT02287896/SAP_003.pdf